CLINICAL TRIAL: NCT01778426
Title: Post-reimbursement Study to Follow Spinal Neurostimulator Devices for Pain Therapy
Brief Title: Post-reimbursement Study to Follow Spinal Neurostimulator Devices for Pain Therapy (French SCS Registry)
Acronym: SME
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: 1051
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-05

CONDITIONS: Chronic Pain Syndrome
Keywords: Chronic neuropathic pain syndrome; Spinal Cord Stimulation; Painstim devices; Efficacy; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Medtronic neurostimulator: Patients suffering from chronic neuropathic pain syndrome implanted (first implant or replacements) with a Medtronic neurostimulator.

SUMMARY:
Observational study to evaluate the long term efficacy of Spinal Cord Stimulation (SCS) over 2 years following SCS implant.

This study is requested by French Health Authorities for reimbursement renewal, to maintain reimbursement for SCS in approved indication in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for Spinal Cord Stimulation (pain therapy)
* Patient implanted for less than 3 months or hospitalized for the implant of a Medtronic neurostimulator including:
* primary implant with Spinal Cord Stimulation indication and positive test of stimulation or
* device replacement of a Medtronic neurostimulator used for Pain Therapy
* Evaluation of usual pain in the back, upper and lower limbs using a visual analogic scale must be available for the 3 days preceding implant.
* Treatments must also be available
* Patient read and signed the data release form

Exclusion Criteria:

* Patient declined participation
* Patient is not available for follow up
* Stimulation of other body part than spinal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients implanted (first implant or replacements) with a Medtronic neurostimulator in selected French sites .
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine DJIAN, MD, Study Chair — Hôpital Saint Anne, Paris
Locations (1):
- Hôpital Foch - 40 rue Worth, Suresnes, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled in the study on January 13, 2012. The last subject was enrolled on December 19, 2013 and the last visit of the last subject was on January 11, 2016. A total of 414 patients were assessed for eligibility, across 28 sites in France, of which, 402 subjects were included in the final analysis.
Pre-assignment Details: Not applicable; this study was non-randomized in which no treatment group was assigned.
Groups:
- Primo-implant (PI): Subjects implanted for the first time with Medtronic SCS devices, in order to assess the effectiveness of the treatment compared to pre-operative situation.
- Replacement (RP): Subjects implanted with a new Medtronic SCS neurostimulator as a replacement of their Medtronic SCS devices, in order to document the integrality of the practice and collect long-term data like complications and definitive explants.
Period: Overall Study - Full Analysis Set (FAS)
Arm/Group | Primo-implant (PI) | Replacement (RP)
Started (Patients included in the study.) | 264 | 138
Completed (Patients having completed the 2 year follow-up.) | 208 | 113
Not Completed | 56 | 25
Period: Intention-To-Treat (ITT) - Completer
Arm/Group | Primo-implant (PI) | Replacement (RP)
Started (Primo-implanted patients with baseline and follow-up pain intensity data at 2 years completed.) | 198 | 0 (Not applicable: ITT-completer contains only primo-implant subjects.)
Completed (Patients having completed the 2 year follow-up.) | 198 | 0 (Not applicable: ITT-completer contains only primo-implant subjects.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS includes all subjects from primo-implant (n=264) and replacement (n=138) groups enrolled in the study with a valid Patient Data Release Form. 402 subjects were analyzed in the FAS.
Groups:
- Primo-implant (PI): Subjects implanted for the first time (primary implant group) with Medtronic SCS devices, in order to assess the effectiveness of the treatment compared to pre-operative situation.
- Replacement (RP): Subjects implanted with a new Medtronic SCS neurostimulator as a replacement of their Medtronic SCS devices (replacement group), in order to document the integrality of the practice and collect long-term data like complications and definitive explants.
- Total: Total of all reporting groups
Arm/Group | Primo-implant (PI) | Replacement (RP) | Total
Number analyzed (Participants) | 264 | 138 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (9.6) | 56.5 (11.4) | 52.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 60 | 177
  Male | 147 | 78 | 225

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least 50% Pain Relief in the Area of Predominant Pain at 2 Years
Description: Percentage of primo-implanted subjects who responded to the treatment, where response was defined as a pain relief of at least 50% in the area with predominant pain intensity from baseline to two years follow-up. Pain intensity was assessed using an 11-point (0-10) Numeric Pain Rating Scale (NPRS) ranging from 0 (no pain) to 10 (maximum pain possible).
Time Frame: 2 years
Population: ITT - completer (n=198) consists of all primo-implant subjects with baseline and follow-up pain intensity data at 2 years completed. Among 198 subjects, 179 patients had a visit at one year completed.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Groups:
- Primo-implant (PI): Subjects implanted for the first time with Medtronic SCS devices
Arm/Group | Primo-implant (PI)
Number analyzed (Participants) | 198
Percentage of responders | 59.1 [51.9 to 66.0]

2. Secondary Outcome: Percentage of Subjects With at Least 50% Pain Relief in the Area of Non-predominant Pain
Description: Percentage of primo-implanted subjects who responded to the treatment, where response was defined as a pain relief of at least 50% in the area with non-predominant pain intensity at 1 and 2 years follow-up, compared to baseline. Pain intensity was assessed using an 11-point (0-10) Numeric Pain Rating Scale (NPRS) ranging from 0 (no pain) to 10 (maximum pain possible).
Time Frame: 1 year and 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Primo-implant (PI)
Number analyzed (Participants) | 198
Percentage of responders
  1 year: number analyzed (Participants) | 130
  1 year | 46.9 [38.3 to 55.5]
  2 years: number analyzed (Participants) | 142
  2 years | 46.5 [38.3 to 54.7]

3. Secondary Outcome: Percentage of Subjects With at Least 50% Pain Relief in the Area of Predominant Pain at 1 Year
Description: Percentage of primo-implanted subjects who responded to the treatment, where response was defined as a pain relief of at least 50% in the area with predominant pain intensity from baseline to one year follow-up. Pain intensity was assessed using an 11-point (0-10) Numeric Pain Rating Scale (NPRS) ranging from 0 (no pain) to 10 (maximum pain possible).
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Primo-implant (PI)
Number analyzed (Participants) | 179
Percentage of responders | 60.7 [53.1 to 67.9]

4. Secondary Outcome: Concomitant Pain Relief Medication
Description: Percentage of primo-implanted subjects taking pain relief medication at baseline, 1 and 2 years.
Time Frame: Baseline, 1 and 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subject taking drug
Groups:
- Primo-implant - Baseline: Subjects implanted for the first time with Medtronic SCS devices. Results at baseline.
- Primo-implant - 1 Year: Subjects implanted for the first time with Medtronic SCS devices. Results at 1 year follow-up.
- Primo-implant - 2 Years: Subjects implanted for the first time with Medtronic SCS devices. Results at 2 years follow-up.
Arm/Group | Primo-implant - Baseline | Primo-implant - 1 Year | Primo-implant - 2 Years
Number analyzed (Participants) | 198 | 179 | 198
Percentage of subject taking drug
  Analgesic, level 1 | 59.1 [51.9 to 66.0] | 43.3 [35.9 to 50.9] | 43.9 [36.9 to 51.2]
  Analgesic, level 2 | 61.1 [53.9 to 67.9] | 35.4 [28.4 to 42.9] | 36.4 [29.7 to 43.5]
  Analgesic, level 3 | 44.9 [37.9 to 52.2] | 19.7 [14.1 to 26.3] | 18.7 [13.5 to 24.8]
  NSAID | 28.8 [22.6 to 35.6] | 9.0 [5.2 to 14.2] | 8.6 [5.1 to 13.5]
  Antiepileptic | 69.7 [62.8 to 76.0] | 38.2 [31.0 to 45.8] | 30.3 [24.0 to 37.2]
  Antidepressant | 54.0 [46.8 to 61.1] | 33.7 [26.8 to 41.2] | 29.8 [23.5 to 36.7]

5. Secondary Outcome: Dose of Analgesics Level 3 (Morphinics)
Description: Dose of analgesics level 3 (morphinics) summarized as equivalent morphine dose at baseline, 1 and 2 years.
Time Frame: Baseline, 1 and 2 years
Population: ITT - completer (n=198) consists of all primo-implant subjects with baseline and follow-up pain intensity data at 2 years completed. Among 198 subjects, 179 patients had a visit at one year completed.
  Here, patients taking analgesics level 3 medications were considered.
Measure: Mean (Standard Deviation); unit: Daily equivalent morphine dose in mg
Arm/Group | Primo-implant - Baseline | Primo-implant - 1 Year | Primo-implant - 2 Years
Number analyzed (Participants) | 89 | 35 | 37
Daily equivalent morphine dose in mg | 90.2 (67.3) | 102.6 (95.8) | 100.3 (94.2)

6. Secondary Outcome: Patient Satisfaction
Description: Percentage of primo-implanted subjects satisfied with the treatment 1 and 2 years after implantation (defined as indicating "pain relief improvement," "daily life improvement," "rather satisfied with the treatment," or "would agree to the treatment again").
Time Frame: 1 and 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects satisfied
Arm/Group | Primo-implant - 1 Year | Primo-implant - 2 Years
Number analyzed (Participants) | 179 | 198
Percentage of subjects satisfied
  Pain relief improvement | 89.9 [84.5 to 93.9] | 89.3 [84.2 to 93.3]
  daily life activity improvement | 82.0 [75.6 to 87.4] | 81.8 [75.7 to 86.9]
  treatment satisfaction | 89.9 [84.5 to 93.9] | 91.4 [86.6 to 94.9]
  agree to the treatment again | 92.1 [87.2 to 95.6] | 92.9 [88.4 to 96.1]

7. Secondary Outcome: Return to Work
Description: Percentage of subjects being invalid at inclusion and active at 1 and 2 years.
Time Frame: 1 and 2 years
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Primo-implant - 1 Year | Primo-implant - 2 Years
Number analyzed (Participants) | 179 | 198
Percentage of subjects | 8 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through the study end.
Description: Adverse events related to the device or procedure (including definitive explant or repositioning) were collected. Whether an event met the criteria of serious was determined by the study site.
Groups:
- Full Analysis Set (FAS): FAS includes all subjects from primo-implant (n=264) and replacement (n=138) groups enrolled in the study with a valid Patient Data Release Form. 402 subjects were analyzed in the FAS.
Arm/Group | Full Analysis Set (FAS)
Serious Adverse Events (participants affected / at risk) | 89/402
Other Adverse Events (participants affected / at risk) | 105/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Analysis Set (FAS) (N=402)
Implant site infection (Infections and infestations) | 8
Peritonitis (Infections and infestations) | 1
Completed suicide (Psychiatric disorders) | 2
Allodynia (Nervous system disorders) | 3
Intercostal neuralgia (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 1
Phantom pain (Nervous system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Death (General disorders) | 1
Device battery issue (General disorders) | 4
Device dislocation (General disorders) | 4
Device end of service (General disorders) | 2
Device extension damage (General disorders) | 1
Device issue (General disorders) | 1
Device lead damage (General disorders) | 1
Device lead issue (General disorders) | 3
Device stimulation issue (General disorders) | 7
Implant site hyperaesthesia (General disorders) | 1
Implant site inflammation (General disorders) | 1
Implant site pain (General disorders) | 7
Medical device discomfort (General disorders) | 1
Medical device site pain (General disorders) | 2
Pain (General disorders) | 30
Surgical skin tear (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Medical device removal (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Analysis Set (FAS) (N=402)
Implant site infection (Infections and infestations) | 7
Infection (Infections and infestations) | 1
Hypersensitivity (Immune system disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Burning sensation (Nervous system disorders) | 2
Meningocele acquired (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 7
Sciatica (Nervous system disorders) | 2
Spinal claudication (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Implant site haematoma (Vascular disorders) | 1
Subcutaneous hematoma (Vascular disorders) | 1
Syncope (Vascular disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Device dislocation (General disorders) | 8
Device ineffective (General disorders) | 2
Device intolerance (General disorders) | 1
Device stimulation issue (General disorders) | 13
Implant site discolouration (General disorders) | 1
Implant site hematoma (General disorders) | 3
Implant site pain (General disorders) | 21
Lead dislodgement (General disorders) | 1
Medical device discomfort (General disorders) | 4
Necrosis (General disorders) | 1
Pain (General disorders) | 29
Therapeutic product ineffective (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Neurostimulator removal (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
The targeted pain area of the therapy was assumed to be the one with the predominant NPRS score at baseline. For the replacement group it was unknown if the therapy was active at the time of the device replacement (enrollment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is stated in the CIP and Agreement signed by the investigators that the French SCS Registry data are the sole property of Medtronic.